CLINICAL TRIAL: NCT04469621
Title: A Phase 1b, Randomized, Double-blinded, Placebo-controlled Study to Evaluate the Safety and Immunomodulatory Effect of the RIPK1 Inhibitor SAR443122 in Hospitalized Patients With Severe COVID-19
Brief Title: A Phase 1b Trial to Evaluate Safety and Effect of SAR443122 on Immune System in Severe COVID-19
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PDY16879; 2020-002104-39 (EudraCT Number); U1111-1250-1185 (Other: UTN)
Record Dates: First submitted 2020-06-28; First posted 2020-07-14 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Corona Virus Infection
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SAR443122 (Experimental): SAR443122 dose 1, twice daily for 14 days
  Interventions: Drug: SAR443122
- Placebo (Placebo Comparator): matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SAR443122 — Pharmaceutical form:capsule Route of administration: oral
  Arms: SAR443122
Drug: Placebo — Pharmaceutical form:capsule Route of administration: oral
  Arms: Placebo

SUMMARY:
Primary Objective:

To evaluate the effect of SAR443122 relative to the control arm on the hyperinflammatory state as measured by C-reactive protein (CRP) levels in adult patients hospitalized with severe coronavirus disease 2019 (COVID-19)

Secondary Objectives:

* To evaluate the time to onset of effect of SAR443122 relative to the control arm on the hyperinflammatory state as measured by CRP levels
* To evaluate the time to onset of effect of SAR443122 relative to the control arm on oxygenation status
* To evaluate the effect of SAR443122 relative to the control arm on oxygenation status
* To evaluate the effect of SAR443122 relative to the control arm on total duration of supplemental oxygen requirement
* To evaluate the effect of SAR443122 relative to the control arm on length of ventilator support needed
* To evaluate the effect of SAR443122 relative to the control arm on laboratory markers of severe COVID-19
* To evaluate the effect of SAR443122 relative to the control arm on mortality
* To evaluate the effect of SAR443122 relative to the control arm on need for thrombolytic therapy
* To evaluate the effect of SAR443122 relative to the control arm on need for vasopressor treatment
* To evaluate the safety of SAR443122 as compared to the control arm up to End of Study
* To evaluate the effect of SAR443122 relative to the control arm on total duration without high flow supplemental oxygen requirements

DETAILED DESCRIPTION:
Study duration per participant is approximatively 32 days including a 14-day treatment period

ELIGIBILITY:
Inclusion criteria:

* Participant must be ≥18 years and ≤80 years of age inclusive, at the time of signing the informed consent.
* Hospitalized (or documentation of a plan to admit to the hospital if the participant is in an emergency department) with evidence of COVID-19 lung disease diagnosed by chest radiograph, chest computed tomography or chest auscultation (rales, crackles) and with severe disease defined as follows: The participant requires supplemental oxygen administered by nasal cannula, simple face mask, or other similar oxygen delivery device (ie, increase in oxygen requirement following SARS-CoV-2 infection).
* SARS-CoV-2 infection confirmed by RT-PCR, or other commercial or public health assay in any specimen, within 3 weeks prior to randomization, and no alternative explanation for current clinical condition.
* At time of randomization, have demonstrated laboratory signs consistent with systemic inflammation.
* Male and/or female participants, including women of childbearing potential (WOCBP).
* Capable of giving signed informed consent.

Exclusion criteria:

* In the opinion of the investigator, unlikely to survive after 48 hours, or unlikely to remain at the investigational site beyond 48 hours
* Participants requiring use of invasive or non-invasive positive pressure ventilation at randomization.
* Presence of significant liver enzyme abnormalities, thrombocytopenia or anemia at screening.
* Any prior or concurrent use or plans to receive during the study period of immunomodulatory therapies (other than interventional drug) at screening.
* Use of chronic systemic corticosteroids for a non-COVID-19-related condition in a dose higher than prednisone 10 mg or equivalent per day at screening.
* Exclusion criteria related to tuberculosis (TB) and non-tuberculous mycobacterial (NTM) infections.
* Participants with suspected or known active systemic bacterial or fungal infections within 4 weeks of screening.
* Pregnant or breastfeeding women.
* In the opinion of the study investigator, might confound the results of the study or pose an undue risk to the safety of the participant.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2020-07-17 (Actual); Primary Completion 2020-10-23 (Actual); Study Completion 2020-10-23 (Actual)

PRIMARY OUTCOMES:
Relative change from baseline in CRP level | Day 7
  Relative change from baseline in CRP level on Day 7

SECONDARY OUTCOMES:
Time to 50% decrease from baseline in CRP level | Baseline to Day 28
  The time to 50% decrease from baseline in CRP level
Time to improvement of oxygenation | Baseline to Day 28
  The time to improvement of oxygenation as measured by oxygen saturation >/=92% breathing room air over 48 hrs or until discharge
Change from baseline in SPO2/FiO2 ratio | Day 7
  Change from baseline in SPO2/FiO2 ratio at Day 7
Number of Days without need for oxygen support and alive | Baseline to Day 28
  Number of Days without need for oxygen support and alive (oxygen saturation >=92% breathing room air) up to Day 28
Numbers of Ventilator-free days and alive | Baseline to Day 28
  Numbers of Ventilator-free days and alive up to Day 28
Change from baseline in markers of inflammation: white blood cell count and differential blood lymphocytes | Day 7 and Day 15
  Change from baseline in white blood cell count and differential blood lymphocytes at Day 7 and End of treatment (EOT)
Change from baseline in marker of inflammation: neutrophil to lymphocyte ratio | Day 7 and Day 15
  Change from baseline in neutrophil to lymphocyte ratio at Day 7 and EOT
Change from baseline in marker of inflammation: interleukin 6 (IL-6) | Day 7 and Day 15
  Change from baseline in IL-6 at Day 7 and EOT
Change from baseline in D-Dimer | Day 7 and Day 15
  Change from baseline in D-Dimer at Day 7 and EOT
Incidence of Deaths | Baseline to Day 28
  Incidence of Deaths up to Day 28
Percentage of participants receiving thrombolytic treatment | Baseline to Day 28
  Percentage of participants receiving thrombolytic treatment up to Day 28
Percentage of participants receiving vasopressor treatment | Baseline to Day 28
  Percentage of participants receiving vasopressor treatment up to Day 28
Incidence of serious adverse events (SAEs), adverse events of special interest (AESI) and treatment-emergent adverse events (TEAEs) leading to treatment discontinuation | Baseline to Day 28
Incidence of TEAEs leading to study discontinuation (primary reason) | Baseline to Day 28
Numbers of Respiratory Failure-Free Days (RFFD) and alive | Baseline to Day 28
  Numbers of Respiratory Failure-Free Days (RFFD) and alive up to Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (10):
- Investigational Site Number 0320001, Caba, Argentina
- Brazil (3):
  - Investigational Site Number 0760003, Porto Alegre
  - Investigational Site Number 0760001, São José do Rio Preto
  - Investigational Site Number 0760002, São Paulo
- Chile (3):
  - Investigational Site Number 1520001, Santiago
  - Investigational Site Number 1520003, Santiago
  - Investigational Site Number 1520002, Talca
- Investigational Site Number 4840001, Monterrey, Mexico
- Russia (2):
  - Investigational Site Number 6430001, Moscow
  - Investigational Site Number 6430002, Moscow

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Clot PF, Farenc C, Suratt BT, Krahnke T, Tardat A, Florian P, Pomponio R, Patel N, Wiekowski M, Lin Y, Terrier B, Staudinger H. Immunomodulatory and clinical effects of receptor-interacting protein kinase 1 (RIPK1) inhibitor eclitasertib (SAR443122) in patients with severe COVID-19: a phase 1b, randomized, double-blinded, placebo-controlled study. Respir Res. 2024 Feb 28;25(1):107. doi: 10.1186/s12931-024-02670-z. PMID 38419035
- See also: PDY16879 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25318&tenant=MT_SNY_9011